CLINICAL TRIAL: NCT06366737
Title: Effectiveness Of Lingual Retractor Versus Clear Aligner Appliances In En-mass Retraction Of Maxillary Anterior Teeth Segment In Adult Patients: A Randomized Clinical Trial
Brief Title: En-mass Retraction by KILBON Versus CAT Appliances
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab mohamed, Principal investigator, PhD candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2024-03-02
Record Dates: First submitted 2024-03-28; First posted 2024-04-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Maxillary Prognathism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KILBON appliance (Active Comparator): en-mass retraction by lingual retractor
  Interventions: Device: KILBON Appliance
- CAT appliance (Active Comparator): en-mass retraction by clear aligner
  Interventions: Device: CAT appliance

INTERVENTIONS:
Device: KILBON Appliance — palatal TAD assissted lingual appliance for en-mass retraction
  Arms: KILBON appliance
Device: CAT appliance — palatal TAD assissted clear aligner
  Arms: CAT appliance

SUMMARY:
en-mass retraction by lingual retractor versus clear alighner therapy

DETAILED DESCRIPTION:
Comparative Effectiveness Of Lingual Retractor Versus Clear Aligner Appliances In Adult Patients With Maxillary Dentoalveolar Protrusion Treated By Upper First Premolars Extraction And Enmass Retraction Of Maxillary Anterior Teeth Segment Using Palatal Orthodontic Miniscrews :A Randomized Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* adult patients with maxillary dentoalveolar protrusion with mild crowding

Exclusion Criteria:

* - adult patients with maxillary dentoalveolar protrusion with moderate to severe crowding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction during & after phase I treatment. | 6 months
  questionnaire

SECONDARY OUTCOMES:
inclination of upper anterior teeth | 6 months
  angle measurement of long axis of maxillary central to maxillary plane in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided